CLINICAL TRIAL: NCT02334917
Title: Comparison of Fast-Absorbing Sutures for Mohs Surgery Repair on the Face (ComFAS): a Randomized Controlled Split-scar Study
Brief Title: Comparison of Fast-Absorbing Sutures for Mohs Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H14-02604
Record Dates: First submitted 2014-11-17; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Cicatrix
Keywords: Suture Comparison
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Absorbable suture closure (Experimental): Patients will have half of their surgical wound closed using one kind of absorbable superficial sutures, and the other half with a different kind of absorbable superficial suture. Which half receives which suture will be randomly determined.
  Interventions: Procedure: Surgical wound closure with superficial absorbable sutures

INTERVENTIONS:
Procedure: Surgical wound closure with superficial absorbable sutures — Different superficial absorbable sutures will be used in the closure of skin wounds after Mohs surgery. No drugs or devices are being compared, only the two different absorbable sutures (Vicryl Rapide and Fast Absorbing Gut).

SUMMARY:
This study is being carried out to assess equivalence of scar outcome for two absorbable sutures used for wound closure on the face in dermatologic surgery: rapidly absorbable polyglactin 910 (VicrylRapide™) and fast-absorbing plain gut (5-0 fast). This is important because absorbable sutures are commonly used in Mohs surgery for epidermal closure, yet there is no evidence indicating if any of the sutures above allow for a better cosmetic outcome (less erythema, edema, and scarring).

DETAILED DESCRIPTION:
Prospective randomized controlled split-scar observer-blinded study.

After dermatologic surgery on the face, surgeons have a choice between using non-absorbable or absorbable sutures for skin closure. A dermatologic surgeon favoring absorbable sutures for wound closure will consider many factors in material selection, including ease of manipulation, cost, and absorption time. However, there have been no randomized trials comparing the most important measure: aesthetic/cosmetic outcome.

Study endpoint/outcome: use three validated scar assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 18 years and are having Mohs surgery on the face.

Exclusion Criteria:

* Patients with surgical wounds less than 4cm in length
* Patients requiring full thickness skin grafts for reconstruction
* Patients who are unable to attend routine postoperative follow-up appointments
* Patients who are receiving radiation therapy after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The Stony Brook Scar Evaluation Scale (SBSES) score (cosmetic outcome) | 6 months
  In this study we will use three validated scar assessment tools (the Stony Brook Scar Evaluation Scale (SBSES) to assess scar width, height, color, cross-hatching and overall appearance, the Wound Evaluation Scale (WES) to rate scar stepoff, contour irregularity, scar width, edge inversion, and inflammation , and the Visual Analogue Scale (VAS)) to assess overall scar appearance. This will be done at the one-week, two-month and six-month post-operative follow-ups.
The Wound Evaluation Scale (WES) score (cosmetic outcome) | 6 months
  In this study we will use three validated scar assessment tools (the Stony Brook Scar Evaluation Scale (SBSES) to assess scar width, height, color, cross-hatching and overall appearance, the Wound Evaluation Scale (WES) to rate scar stepoff, contour irregularity, scar width, edge inversion, and inflammation , and the Visual Analogue Scale (VAS)) to assess overall scar appearance. This will be done at the one-week, two-month and six-month post-operative follow-ups.
The Visual Analogue Scale (VAS) score (cosmetic outcome) | 6 months
  In this study we will use three validated scar assessment tools (the Stony Brook Scar Evaluation Scale (SBSES) to assess scar width, height, color, cross-hatching and overall appearance, the Wound Evaluation Scale (WES) to rate scar stepoff, contour irregularity, scar width, edge inversion, and inflammation , and the Visual Analogue Scale (VAS)) to assess overall scar appearance. This will be done at the one-week, two-month and six-month post-operative follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: David M Zloty, MD, Principal Investigator — University of British Columbia